CLINICAL TRIAL: NCT07063173
Title: Bioavailability of Ration Items Containing Tart Cherry Extract
Acronym: Tart Cherry
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 24-07
Record Dates: First submitted 2025-03-17; First posted 2025-07-14 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Bioavailability
Keywords: military; tart cherry; muscle recovery; polyphenols

STUDY DESIGN:
Intervention Model Description: In this randomized, crossover study, participants will consume three different food products containing TC component and a control (food item without TC) over four different sessions. Each session will be followed by a five-day washout period.
Masking Description: One of four test food items will be consumed on the morning of each test trial (randomly assigned).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tart Cherry Juice (Active Comparator): The commercially available tart cherry (TC) drink contains 100% concentrated Montmorency cherry juice (CherryActive, Sunbury, UK) as a "gold standard". Participants will consume 60 mL of the concentrate diluted with 500 mL of water, which delivers ~120 mg of anthocyanins.
  Interventions: Dietary Supplement: Fruit Bar; Dietary Supplement: Powdered Drink; Dietary Supplement: Placebo beverage
- Fruit Bar (Active Comparator): The fruit powder is incorporated into a snack bar, which delivers ~120 mg of anthocyanins.
  Interventions: Dietary Supplement: Powdered Drink; Dietary Supplement: Commercially available 100% tart cherry juice; Dietary Supplement: Placebo beverage
- Powdered Drink (Active Comparator): The fruit powder is incorporated into a powdered drink, which delivers ~120 mg of anthocyanins..
  Interventions: Dietary Supplement: Fruit Bar; Dietary Supplement: Commercially available 100% tart cherry juice; Dietary Supplement: Placebo beverage
- Control Beverage (Placebo Comparator): A control powdered drink will be formulated with similar organoleptic qualities to the TCP-containing powdered drink without containing any polyphenol-rich ingredients.
  Interventions: Dietary Supplement: Fruit Bar; Dietary Supplement: Powdered Drink; Dietary Supplement: Commercially available 100% tart cherry juice

INTERVENTIONS:
Dietary Supplement: Fruit Bar — Tart Cherry N185
  Other Names: Tart Cherry N185
  Arms: Control Beverage; Powdered Drink; Tart Cherry Juice
Dietary Supplement: Powdered Drink — Vita Cherry Sport N1244 (FutureCeuticals, Momence, IL)
  Other Names: Vita Cherry Sport N1244
  Arms: Control Beverage; Fruit Bar; Tart Cherry Juice
Dietary Supplement: Commercially available 100% tart cherry juice — 100% concentrated Montmorency cherry juice (CherryActive, Sunbury, UK)
  Other Names: "gold standard" beverage
  Arms: Control Beverage; Fruit Bar; Powdered Drink
Dietary Supplement: Placebo beverage — Placebo beverage
  Arms: Fruit Bar; Powdered Drink; Tart Cherry Juice

SUMMARY:
To determine how consuming food items containing shelf-stored tart cherry impacts your body's ability to absorb and use the compounds within tart cherry.

DETAILED DESCRIPTION:
Consumption of tart cherry (TC) products may have beneficial effects on military performance. For example, in-vitro and in-vivo evidence indicates the benefits of TC products on muscle. This includes reduced muscle damage, muscle soreness and strength decrements after resistance exercise; and increased antioxidant capacity, reduced inflammation and reduced lipid peroxidation following endurance exercise. Prior to assessing potential performance benefits, DEVCOM-Soldier Center's Combat Feeding Division (CFD) is seeking to determine the effect of shelf-stable tart cherry powder (TCP)-containing food items on the bioavailability and absorption of polyphenols in humans.

The primary objective of his study is to evaluate the postprandial concentrations of anthocyanins, anthocyanidins, flavonols, phenolic acids, and their degradation products in response to a TCP-containing, shelf-stable bar and shelf-stable powdered drink, compared to a non-TCP containing control item and a TC-containing commercial item. Secondary objectives are to determine postprandial polyphenol absorption via urine concentrations of anthocyanins, anthocyanidins, flavonols, phenolic acids and their degradation products; and circulating antioxidant capacity. Active-duty military personnel and civilians will be invited to participate in the study if they are between the ages of 18 (or 17 for military personnel) and 39, are willing to participate in all study procedures and comply with all study instruction and pass a general medical clearance.

In this randomized, crossover study, participants will consume three different food products containing TC component and a control (food item without TC) over four different sessions. Each session will be followed by a five-day washout period. On the day of each experimental session, and after verification of compliance with study procedures (e.g., overnight fast and low polyphenol diet day prior…), an IV catheter will be inserted, and an initial blood sample will be collected. Immediately following, volunteers will consume either: 1) commercially available TC juice ("gold standard"), 2) CFD-formulated snack bar containing TCP, 3) CFD-formulated powdered drink containing TCP, or 4) CFD-formulated beverage containing no polyphenols (Figure 1). TC containing treatments will be matched by total anthocyanin content (~120 mg total). Blood samples will be collected on the day of each session and the day after for measurement of circulating phenolic compounds (by CFD using LC-MS). Biomarkers of oxidation and anti-oxidation will also be measured, along with associations between study outcomes and gut microbiome composition. Complete data will be collected for up to 15 participants.

ELIGIBILITY:
Inclusion Criteria:

* Active duty military personnel and civilians will be invited to participate in the study if they:

  * Are between the ages of 18 (or 17 for military personnel) and 39.
  * Are willing to participate in all study procedures and comply with all study instruction.
  * In good health as determined by OMSO (Office of Medical Support and Oversight).
  * Supervisor approval for federal civilian employees and non-HRV active-duty military personnel stationed at NSSC

Exclusion Criteria:

* • Unable to understand verbal or written instructions or testing materials in English.

  * Have a bleeding disorder (e.g., von Willebrand Disease, hemophilia) or are being treated with medication that will impair blood clotting (for example, coumadin)
  * Have a history of GI-related conditions that may impact macronutrient absorption (e.g., Crohn's disease, ulcerative colitis, Celiac's disease or gluten sensitivity, bariatric surgery or gastroparesis, short bowel, inflammatory bowel disease, etc…);
  * Any use of antibiotics or antifungal, except topical antibiotics/antifungals within 3 months of study participation.
  * Colonoscopy within 3 months of study participation.
  * Regular (i.e., weekly or more frequent) use of over-the-counter medications (including antacids, laxatives, stool softeners, and antidiarrheals) unless approved by OMSO and study PI.
  * Are habitually taking nonsteroidal anti-inflammatory drugs (e.g., Advil, aspirin), corticosteroids (e.g., prednisone) or immunosuppressants (e.g. Humira);
  * Have an allergy or aversion (extreme dislike) to any of the test foods(e.g., cherry flavored beverages or bar). Allergy symptoms may include anaphylaxis, hives or eczema, tingling/itching in the mouth, dizziness or fainting, diarrhea, nausea or vomiting, swelling of the lips, face, tongue and throat).
  * Have donated blood within the past 8 weeks of the first test session or plan to donate blood during the study.
  * Are not willing to abstain from tobacco products and vigorous exercise for at least 24 hours" before each trial and consume a low-polyphenol diet two days prior to each test session and on the day of the test session.

Ages: 17 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Postprandial concentrations of polyphenols in plasma | Baseline and postprandially @ 30-minutes, 60-minutes, 120-minutes, 240-minutes, 360-mins, 24 hours
  The primary objective of this study is to evaluate the postprandial concentrations of:
  * nmol/L for anthocyanins & anthocyanidins (cyanidin-3-glucosylrutinoside, cyanidin-3-rutinoside,cyanidin-3-sophoroside, cyanidin-3-glucoside, cyanidin, peonidin-3-glucoside and pelargonidin);
  * µmol/L for flavonols (Isorhamnetin-3-rutinoside, kaemperol, and que after consuming a TCP-containing, shelf-stable bar and shelf-stable powdered drink (compared to a non-TCP containing control and a TC-containing commercial item).

SECONDARY OUTCOMES:
Postprandial concentrations of polyphenols in urine | Baseline and postprandially @ Baseline and postprandially @ 30-minutes, 60-minutes, 120-minutes, 240-minutes, 360-mins, 24 hours
  Secondary objectives are to determine postprandial polyphenol absorption via urine concentrations of anthocyanins, anthocyanidins, flavonols, phenolic acids and their degradation products as well as circulating antioxidant capacity; and to determine associations between these outcomes and gut microbiome composition

CONTACTS AND LOCATIONS:
Overall Officials: Tracey Smith, PhD, Principal Investigator — United States Army Research Institute of Environmental Medicine
Locations (1):
- USARIEM, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
The principal investigator, with the assistance of associate investigators and project coordinator, will continuously evaluate recruitment, the informed consent process, adverse events, and protocol adherence and deviations in order to identify unanticipated problems or risks to the participants associated with the research. The principal investigator will ensure that the number of participants recruited for this study complies with the protocol. The principal investigator will be responsible for continually monitoring that data for each participant is collected and analyzed as specified in this protocol, and for ensuring that study files and IRB documentation are appropriate and up to date. The principal investigator and OMSO staff will discuss "discontinuation criteria" for individual participants as the study progresses, based on their observations of the participant during testing or non-testing periods.

DOCUMENTS (1):
  • Informed Consent Form (2024-03-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT07063173/ICF_000.pdf